CLINICAL TRIAL: NCT00471861
Title: Does Migraine As A Partly Inflammatory Disease Increase The Inflammatory Markers Of The Patient When Actively Having a Migraine?
Brief Title: Inflammatory Markers in Patients With Active Migraine Headaches
Status: Completed | Type: Observational
Sponsor: Westside Family Medical Center, P.C. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Gary E. Ruoff, Westside Family Medical Center
Other Study IDs: 109944
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2009-02

CONDITIONS: Migraine
Keywords: Inflammatory Markers; Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether C-Reactive Protein (CRP) is elevated in patients with active migraine headaches. Secondary goal is to determine whether other inflammatory markers, such as Calcitonin Gene Peptide (CGRP), Vasoactive Intestinal Polypeptide (VIP) or Substance P (SP) are elevated in patients having a migraine headache.

DETAILED DESCRIPTION:
A random selection of patients both male and female from a primary care practice with a diagnosis of having migraine headaches will be enrolled. Thirty (30) patients will be recruited mainly from the primary care practice. Recruitment will include males and females aged 21-65. The patients who meet the inclusion criteria will be enrolled. The patients who do not have migraine headaches will also be enrolled and function as controls. Non-migraine patients will meet inclusion criteria 1, 2 and 3 and all of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign a written informed consent.
2. Enrollment population would include males and females 21 years of age to 65 years of age.
3. Non-migraine subjects will be allowed in the control group
4. Have episodic migraine headaches
5. Patients to satisfy the diagnosis of migraine headaches with aura, without aura or mixed.
6. Must be able to differentiate migraine headaches from other headaches

Exclusion Criteria:

1. Any medical condition in the opinion of the investigator that would make the subject unsuitable for enrollment.
2. Basilar or hemiplegic migraine headaches.
3. Pregnant woman or a nursing mother
4. History (within 1 year) or current evidence of drug or alcohol abuse.
5. More than 15 migraine headaches per month
6. Chronic daily headaches
7. Chronic use of NSAIDs
8. Current participation in a research study or within the last 30 days.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migraine
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-05; Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Ruoff, MD, Principal Investigator — Westside Family Medical Center, P.C.
Locations (1):
- Westside Family Medical Center, P.C., Kalamazoo, Michigan, United States